CLINICAL TRIAL: NCT05642182
Title: A Study of Improvement in Psoriasis Symptoms Associated with Combinations of Biologically Active Natural Substances (SFA-002) with Known Safety Profile
Brief Title: Study of SFA002 in Patients with Mild to Moderate Psoriasis Plaques
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SFA Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SFA002-002
Record Dates: First submitted 2022-05-03; First posted 2022-12-08 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Psoriasis
Keywords: Mild Plaques psoriais; moderate Plaque Psoriasis; Severe plaque psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug (SFA002) Formula 1 (Experimental)
  Interventions: Drug: SFA002
- Drug (SFA002) Formula 2 (Experimental)
  Interventions: Drug: SFA002

INTERVENTIONS:
Drug: SFA002 — Study drug formula without excipient
  Arms: Drug (SFA002) Formula 1
Drug: SFA002 — Study Drug SFA002 with excipient (Propionate)
  Arms: Drug (SFA002) Formula 2

SUMMARY:
The purpose of this study is to determine the safety, metabolism and potential effect of drug product SFA-002 on mild moderate and severe chronic plaque psoriasis. Psoriasis is a common chronic skin disorder that affects over 4 million people. There is no cure for psoriasis and treatment is directed at controlling patients' symptoms.

DETAILED DESCRIPTION:
Up to ninety volunteers with mild to moderate chronic plaque psoriasis will be recruited for an open label 24 week prospective study of the safety of 2 different dosages for 12 weeks of active therapy and 12 weeks of follow up. Blood will be drawn to determine any clinical effect on each group at the 12 week time mark and residual effects after 24 weeks. Throughout the study the investigators will perform both clinical and laboratory assessments to measure safety and response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes ≥18 years of age with at least one skin plaque that is >5 cm2 due to known psoriasis considered clinically to be MILD to MODERATE or MODERATE to SEVERE during evaluation and diagnosis at least 1 year prior. Mild is defined as "Just detectable to mild thickening; pink to light red coloration; predominantly fine scaling", whereas moderate is defined as "Clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling".
* Have or have not been treated with phototherapy, systemic therapy, or other therapies for their psoriasis
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use effective contraceptive methods (such as abstinence, intrauterine device (IUD), or double barrier device) during the study and for at least 3 months following completion of the study.
* Mentally competent, able to understand and willingness to sign the Informed Consent Form (ICF).
* Able to undergo the investigations and to follow the visit schedule stated in the study protocol.

Exclusion Criteria:

* The forms of psoriasis other than chronic plaque psoriasis (such as drug-induced psoriasis or guttate, erythrodermic, or pustular psoriasis) or if the psoriasis does not meet the criterion of chronicity (defined as a clinically significant flare of psoriasis within 12 weeks before baseline).
* Presence of other form of inflammatory skin diseases (such as atopic dermatitis) or infectious diseases (such as cellulitis, warts, fungal cutaneous diseases, etc.)
* A clinically significant flare of psoriasis within 12 weeks before baseline. (Note: The determination of whether prospective study participants had a "significant flare" prior to study baseline is left to the investigators. The intent of this criterion was to ensure the condition is sufficiently stable and aligned with the chronic nature of plaque psoriasis, so that an adequate assessment of the efficacy could be made.)
* Prior or current use of psoriasis medications that might confound assessment of efficacy of the investigational supplements used in this study, unless there were used before their washout period prior to study initiation (see Table 2 for specific medications and their washout periods).
* Known serious medical illness, such as significant cardiac disease (e.g., symptomatic congestive heart failure, unstable angina pectoris, symptomatic coronary artery disease, myocardial infarction within the past 6 months, uncontrolled or symptomatic cardiac arrhythmia, or New York Heart Association Class III or IV), or severe debilitating pulmonary disease, that would potentially increase subjects' risk for toxicity.
* Known to have a history of risk factors for torsade de pointes (e.g., clinically significant heart failure, hypokalemia, family history of Long QT Syndrome).
* Known to have arterial thrombotic event, stroke, or transient ischemia attack within the past 12 months.
* Known to have uncontrolled hypertension (systolic blood pressure >160 mm Hg or diastolic blood pressure >90 mm Hg), or peripheral vascular disease ≥grade 2.
* Known to have active central nervous system (CNS), epidural tumor or metastasis, or brain metastasis.
* Any active uncontrolled bleeding, a bleeding diathesis (e.g., active peptic ulcer disease), or a history of bleeding (e.g., hemoptysis, upper or lower gastrointestinal [GI] bleeding) within the past 6 months.
* Dyspnea with minimal to moderate exertion; large and recurrent pleural or peritoneal effusions requiring frequent drainage (e.g. weekly); or any amount of clinically significant pericardial effusion.
* Diabetes of any type, except Non-Insulin Dependent Diabetes Mellitus (NIDDM) that is controlled and with hemoglobin A1c 8%.
* Evidence of active infection during screening, or serious infection within the past month.
* Patients with known Human Immunodeficiency Virus (HIV), hepatitis B or C virus (HBV) or (HCV), respectively), or active or latent Tuberculosis (TB).
* Serious or non-healing wound, skin ulcer, or bone fracture.
* Abdominal fistula, GI perforation, or intra-abdominal abscess within the past 6 months.
* Neuropathy of grade ≥2.
* Pregnant or lactating females.
* Patients like to purposely undergoing sunlight exposure, including the skin area where the plaques being investigated are located, during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) Score | From enrollment to final visit at 24 weeks treatment and 4 week follow-up
  +/- % Change in Psoriasis (PASI) index from baseline measurement at first dose

SECONDARY OUTCOMES:
Change in IGA score | From enrollment to final visit at 24 weeks treatment and 4 week follow-up
  % Patients achieving 2 point change in IGA Score on 5 point scale and/or score of 2 (almost clear) or 1 Clear.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - NuLine Clinical Trial Center, Pompano Beach, Florida
  - Axis Clincals USA/ Red River Research Patners. LLC, Fargo, North Dakota
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No